CLINICAL TRIAL: NCT06769295
Title: A Phase II Study of AK112 (PD-1/VEGF Bispecific) in Combination with Chemotherapy for Patients with Advanced Non-squamas Non-mall Cell Lung Cancer and Malignant Pleural Effusion
Brief Title: A Phase II Study of AK112 (PD1/VEGF Bispecific) in Combination with Chemotherapy in Patients with NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX-AK112-01
Record Dates: First submitted 2025-01-03; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: NSCLC; AK112; MPE; combination therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- non-Squamous NSCLC with MPE:AK112 plus Chemotherapy (Experimental): non-Squamous NSCLC with malignant pleura effusions:Subjects receive AK112 plus Pemetrexed/Taxol and Carboplatin/Cispaltin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK112 plus Pemetrexed until progression.
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK112 — non-Squamous NSCLC with malignant pleura effusions:Subjects receive AK112 plus Pemetrexed and Carboplatin/Cisplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK112 plus Pemetrexed until progression.
  Other Names: Pemetrexed; Carboplatin/Cisplatin

SUMMARY:
This is a phase II study. All patients are stage IV non-squamas non-small cell lung cancer(NSCLC) with malignant pleura effusion, Eastern Cooperative Oncology Group (ECOG) performance status 0-2. The purpose of this study is to evaluate the efficacy and safety of AK112 in combination with chemotherapy in patients with NSCLC with malignant pleura effusion.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old (at the time of inform consent obtained)；
* Have histologically- or cytologically-confirmed diagnosis of Stage IV non-squamas NSCLC；
* The presence of malignant pleural effusion (positive pleural effusion cytology or multiple pleural nodules or thickening with pleural effusion on CT imaging)；
* Driver gene mutation negative；
* Have a life expectancy of at least 3 months；
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2；
* Has adequate organ function；
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator；
* Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue obtained from either a core or excisional tumor biopsy；
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment；
* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).

Exclusion Criteria:

* Histological or cytological pathology confirmed the presence of small cell carcinoma components, or the main component is squamous cell carcinoma；
* Active malignancies within the past 3 years, with the exception of tumors in this study and cured local tumors；
* Is currently participating in a study of an investigational agent or using an investigational device;
* Active autoimmune disease requiring systemic treatment within 2 years prior to the start of study treatment；
* Subjects who received any prior treatments targeting VEGFR;
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected);
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 12 months prior to day 1 of study treatment;
* Has undergone major surgery within 30 days prior to the first dose of study treatment;
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment NOTE: Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study;
* Has received a live virus vaccine within 30 days prior to first dose of study treatment；

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR of MPE | Up to approximately 2 years
  ORR of malignant pleura effusions is the proportion of subjects with CR or PR , based on WHO Evaluation Criteria .

SECONDARY OUTCOMES:
PFS of MPE | Up to approximately 2 years
  PFS of MPE is defined as the time from the date of randomization till the first documentation of effusion progression (per WHO criteria) assessed by the investigator or death due to any cause (whichever occurs first).
ORR | Up to approximately 2 years
  ORR is the proportion of subjects with CR or PR , based on RECIST v1.1.
PFS | Up to approximately 2 years
  PFS is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
OS rate of 1y | 1 year
  Overall survival rate of 1 year，OS is the time from the date of randomization or first dosing date to death due to any cause.
DOR | Up to approximately 2 years
  DOR is the time between the first observed tumor responseto disease progression or relapse based on RECIST Version 1.1
DCR | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1
OS | Up to approximately 2 years
  OS is the time from the date of randomization or first dosing date to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Wang, Prof, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes